CLINICAL TRIAL: NCT05478915
Title: Outcomes of Surgical Management of Temporomandibular Joint Anterior Disc Displacement Without Reduction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelaal Ali, assistant lecturer of maxillofacial surgery, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-6-12
Record Dates: First submitted 2022-06-22; First posted 2022-07-28 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Temporomandibular Joint Disc Displacement, Without Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with TMJ anterior disc displacement (Experimental): patients had clinically limited mouth opening and by MRI we found anterior disc displacement
  Interventions: Procedure: discectomy of the TMJ disc; Procedure: TMJ discopexy

INTERVENTIONS:
Procedure: discectomy of the TMJ disc — removal of the TMJ disc
Procedure: TMJ discopexy — fixation of the TMJ disc

SUMMARY:
this study will be done to detect the best management of temporo-mandibular joint anterior disc displacement without reduction, for diagnosis, we use MRI on the TMJ to detect status of the disc and joint space, for management, we try to select best operation as discopexy, discectomy with or without replacement, and we follow up the patients and detect side effects and effect for each operation

DETAILED DESCRIPTION:
Discopexy is a procedure in which the displaced disk is freed by the surgeon and lysing adhesions first. The success of the disc repositioning depends on the degree of deformity and the extent of degenerative changes at the time of the arthroplasty. Repositioning the disc restores the condylar movement that was previously blocked by the displaced disc, stabilizes the joint, and improves nutrition and lubrication of articular cartilage. In addition, the workload of the masticatory muscles is reduced when the obstructing disc is repositioned. TMJ disc repositioning surgery seems to improve pain, mouth opening, and patient quality of life

Temporomandibular Joint (TMJ) arthroscopy is one of the most advanced and a minimally invasive technique involving optical instrumentation and prescribed surgical armamentarium, used for the treatment of the TMJ disorders. It is one of the most popular and effective methods of diagnosing and treating TMJ disorders since TMJ disorders have become an increasingly widespread problem in our society. Also, it enables the surgeon to visualize the joint and, therefore, contributes to the diagnosis of the internal pathological condition of the joint and allows inspection of a surgically undisturbed joint both at rest and in function

ELIGIBILITY:
Inclusion Criteria:

* This study will include patients diagnosed as anterior disc displacement without reduction based on clinical manifestations and MRI.

Exclusion Criteria:

* o Patients with severe osteoarthritic changes of the condyle and glenoid fossa.

  * Patients with bony ankylosis.
  * Patients with infection or tumors around joint area.
  * Patients with previous TMJ surgery.
  * Any patient with systemic inflammatory disease or myopathic disease affecting TMJ such as Rheumatoid Arthritis And Systemic Lupus Erythromatosis.
  * Patients unfit for intervention.
  * Patients who refused to share in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-13 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
pain of the TMJ | 6 months
  degree of pain related to TMJ measured by Visual Analogue Scoring System from 0 to 10 where 0 means no pain and 10 means severe unbearable pain

SECONDARY OUTCOMES:
mouth openning | 3 months
  degree of mouth opening measured in centimeters measured by ruler

CONTACTS AND LOCATIONS:
Overall Officials: Kamal M El- sharkawy, proffessor, Study Director — sohag univesity hospitals
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD will be shared with other researchers through NIH(national institute of health)